CLINICAL TRIAL: NCT02704871
Title: To Assess the Performance of SeptiCyte® Lab to Diagnose Patients Identified as Suspected of Sepsis in General Medical and Surgical Wards With Infection-positive From Infection-negative SIRS
Brief Title: The Ward Study for SeptiCyte® Lab to Distinguish Between Infection-positive and Infection-negative SIRS
Status: Terminated | Type: Observational
Why Stopped: Recruitment considerations only and not because of safety or outcomes issues
Sponsor: Immunexpress (Industry)
Collaborators: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IXP 04-01b
Record Dates: First submitted 2016-03-02; First posted 2016-03-10 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Sepsis; SIRS
Keywords: SeptiCyte
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and plasma specimens for nucleic acid and protein analysis
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: SeptiCyte Lab molecular diagnostic test (non-interventional) — This is not an interventional study. Rather it involves evaluation of a molecular diagnostic test to distinguish between sepsis and infection-negative SIRS based on host response.

SUMMARY:
A non-interventional, prospective observational study to assess the performance of SeptiCyte® Lab to diagnose patients identified as suspected of sepsis in general medical and surgical wards with infection-positive from infection-negative SIRS

DETAILED DESCRIPTION:
This study is evaluating a molecular diagnostic device developed to distinguish between sepsis and infection-negative SIRS among critically ill patients.

This study is a prospective, non-randomized, non-interventional, observational trial of patients with suspected sepsis in the medical and/or surgical wards. The study is being conducted on two preselected patient care units.

All patients identified by a local screening tool undergo physician review. If the suspicion of sepsis is found to be plausible, routine and conventional diagnostic procedures, including: routine bloods, blood culture and specialized tests are conducted.

Blood collection for SeptiCyte® Lab and SeptID® is drawn within 6 hours of a positive screen - both use peripheral blood as the clinical sample. The diagnostic performance of the two experimental assays will be compared to Retrospective Physician Diagnosis (RPD), and conventional microbiological culture. The results of SeptiCyte® Lab and SeptID® are not used in any clinical decision-making.

This data will be used to analyze the performance of SeptiCyte® Lab according to the endpoint measures.

ELIGIBILITY:
Inclusion Criteria:

1. 18-89 years old on the day of enrollment.
2. Currently admitted to study designated medical or surgical ward
3. Have a clinical suspicion of sepsis as determined by two physicians after identification by hospital screening tool.
4. Screened positive for sepsis, severe sepsis or septic shock using the RISE2 screening tool.
5. Completed SBAR handover (Situation, Background, Assessment, Recommendation)
6. SIRS present as defined by the presence of two or more of the following:

   * Temperature > 38°C or < 36°C
   * Heart Rate > 90 beat/min
   * Tachypnea > 20/min or PaCO2 < 32 mmHg
   * WBC count > 12 000/mm3 or < 4 000/mm3 or > 10% immature neutrophils (bands)

Exclusion Criteria:

1. Consent not provided
2. Patients less than 18 years of age, or 90 years of age or older.
3. Patients for which a blood sample could not be taken within 24 hours of a physician first determining a clinical suspicion of sepsis.
4. Patients that are not located in the designated medical or surgical ward associated with the study.
5. Patients listed for "Comfort Measures Only".
6. Less than 2 SIRS criteria
7. Commencement of narrow spectrum directed antibiotics prior to screening.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older, previously admitted to medical and/or surgical general hospital wards, who are suspected of sepsis as identified by an in-hospital early-warning screening tool.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
SeptiCyte® Lab test result versus Retrospective Physician Diagnosis (RPD) result | 7 days
  To validate the ability of the SeptiCyte® Lab test to correctly discriminate infection positive from infection negative SIRS in hospital ward patients with two or more SIRS criteria compared to the non-reference method of retrospective physician diagnosis (RPD).

SECONDARY OUTCOMES:
SeptiCyte® Lab test result versus test results for other sepsis biomarkes, including leukocytosis, bandemia, & procalcitonin | 7 days
  To compare SeptiCyte® Lab test scores with other clinical sepsis biomarkers to assess its ability to discriminate infection positive from infection negative SIRS.

OTHER OUTCOMES:
SeptiCyte® Lab test result versus a generalized sepsis screening protocol for identifying potential cases of sepsis | 1 day
  To compare true positive rates of sepsis diagnosis in patients identified only by the RISE2 screening protocol vs. RISE2 screening protocol plus SeptiCyte® Lab results on Day 1.
SeptID® test result versus microbiological reference methods for identifying pathogen(s) | 7 days
  To assess the performance of the SeptID® test against microbiological reference methods for identifying the a pathogen via blood culture.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Levy, MD, Principal Investigator — Rhode Island Hospital; Steven Opal, MD, Principal Investigator — Memorial Hospital of Rhode Island
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available.

REFERENCES:
- See also: Sponsor's website — http://immunexpress.com